CLINICAL TRIAL: NCT01260220
Title: Randomized Trial of Segmental Versus Circumferential Antral Ablation in Paroxysmal Atrial Fibrillation
Acronym: CABLE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Responsible Party: Dr. Lorne J. Gula, Assistant Professor of Medicine, Cardiology, London Health Science Centre
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R-09-489
Record Dates: First submitted 2010-06-08; First posted 2010-12-15 (Estimated); Last update posted 2017-08-28 (Actual); Status verified 2017-08

CONDITIONS: Paroxysmal Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Circumferential (Active Comparator): Completing a complete circle of RF lesions around the left and right pulmonary veins
  Interventions: Procedure: Circumferential Antral Ablation
- Segmental (Experimental): Isolating the left and right pulmonary veins through RF lesions with a segmental antral approach.
  Interventions: Procedure: Segmental Antral ablation

INTERVENTIONS:
Procedure: Circumferential Antral Ablation — The goal is to complete ablation in all segments around the pulmonary veins until a circle of ablation lesions is created in the antrum with at least 30 seconds of ablation, 25W on the posterior surface, 30W on the anterior surface at each site, and change in the local electrogram. Entry and Exit block will be confirmed in each vein. The left superior pulmonary vein and left inferior pulmonary vein will be isolated with one circle, and the right superior and right inferior pulmonary veins will be isolated with one circle.
  Arms: Circumferential
Procedure: Segmental Antral ablation — If the patient is in atrial fibrillation, ablation will begin in the segment with the highest frequency signals in the pulmonary vein antrum. If the patient is in sinus rhythm, mapping and ablation will occur during coronary sinus pacing. Segments with the earliest signals in the Lasso catheter will be targeted, and reassessed after each ablation lesion. This will continue in a segmental fashion on the antrum until pulmonary vein isolation is achieved. Lasso should be moved between veins between lesions to assess the earliest electrogram. Entry and exit block will be confirmed at each vein.
  Arms: Segmental

SUMMARY:
An isolation-limited segmental antral approach to pulmonary vein isolation is as effective in achieving long-term freedom from atrial fibrillation as the standard anatomic, circumferential antral ablation.

DETAILED DESCRIPTION:
This is a randomized controlled non-inferiority designed trial.

Follow up:

Patients will stop their anti-arrhythmic drugs 2 months post procedure. Follow-ups will involve clinical assessment, holter and/or loop recorders at 3, 6, 9, and 12 month intervals.

ELIGIBILITY:
Inclusion Criteria:

* Paroxysmal Atrial Fibrillation (PAF) for at least 6 months with at least 1 symptomatic episode during the previous 6 moths
* Patient must be felt to be candidates for Atrial Fibrillation (AF) ablation based on AF that is symptomatic and refractory or intolerant to at least one class 1 or 3 anti-arrhythmic agent
* Documentation of at least one episode of AF on 12 lead ECG, TTM or Holter monitor within 12 months of randomization in the trial
* Patient must be on continuous anti-coagulation with warfarin (INR 2-3) or fractionated subcutaneous heparin for >4 weeks prior to the ablation or they have undergone a recent (less than 48 hours before planned ablation) transoesphageal echocardiogram to exclude left atrial thrombus.
* Patient must provide written informed consent to participate in the clinical trial

Exclusion Criteria:

* Contraindications to oral anticoagulants
* History of any previous ablation for AF
* Intracardiac thrombus
* AF due to reversible causes
* Pregnancy
* atriotomy scar (typically, MV or TV repair/replacement, ASD surgery, transplants)(CABG are okay)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2009-11-12 (Actual); Primary Completion 2015-12-31 (Actual); Study Completion 2015-12-31 (Actual)

PRIMARY OUTCOMES:
Freedom from atrial fibrillation | six months
  Symptomatic atrial fibrillation recurrence (without anti-arrhythmic med's)

SECONDARY OUTCOMES:
Procedure time | (4-6) hours From the time patient is draped to the time electrophysiology catheters are removed from the body (same day in the electrophysiology lab)
  How long did the procedure take?
Ablation Time | (4-6 hours) Measured during the procedure.
  A cumulative measurement of the duration of ablation used during the pulmonary vein isolation procedure.
Fluoroscopy Time | (4-6 Hours) Measured during the procedure.
  A cumulative measurement of flouroscopy time during the pulmonary vein isolation procedure.
complications | 6 months
  Did the patient experience any complication during the actual pulmonary vein isolation procedure or complication during follow-up related to the procedure?

CONTACTS AND LOCATIONS:
Overall Officials: Lorne J Gula, MD, Principal Investigator — Western University, Canada
Locations (1):
- London Health Science Centre, London, Ontario, Canada